CLINICAL TRIAL: NCT06664437
Title: Efficacy of Adding Neural Mobilization to Joint Mobilization in Patients With Adhesive Capsulitis
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Mohammad Moustafa Aldosoukki Hegazy, Principle investigator, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCBR-353/2024; 2024/03/29095 (Other Grant/Funding Number: Prince Sattam bin Abdulaziz University)
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive capsulitis; Shoulder disability; Joint mobilization
MeSH Terms: conditions — Bursitis | interventions — Exercise; Dosage Forms

STUDY DESIGN:
Intervention Model Description: Interventional procedures:
  Group (A): GH Joint mobilization techniques (Posterior, Inferior glide). Patients were in supine lying position during the whole treatment. The techniques were performed in a rhythmic way, with 2 seconds of glide distraction and then a 2-second break. Each technique was done for 2 minutes [36]. Posterior gliding was performed by maintaining lateral humeral distraction with the glenohumeral in abduction range and the scapula stabilized. Then the therapist applied posterior glide in an oscillating manner. For inferior gliding, with the scapula stabilized, the therapist maintained lateral humeral distraction while applying inferior glide in the resting position of the glenohumeral joint. Patients had 3 sessions of joint mobilization per week for 6 weeks.
  Group (B): Median nerve mobilization techniques (ULLT-1) in addition to GH joint mobilization
  Patients also in this group remained in supine lying position. Median nerve mobilization was performed by placin
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Group (A): GH Joint mobilization techniques (Posterior, Inferior glide). Patients were in supine lying position during the whole treatment. The techniques were performed in a rhythmic way, with 2 seconds of glide distraction and then a 2-second break. Each technique was done for 2 minutes [36]. Posterior gliding was performed by maintaining lateral humeral distraction with the glenohumeral in abduction range and the scapula stabilized. Then the therapist applied posterior glide in an oscillating manner. For inferior gliding, with the scapula stabilized, the therapist maintained lateral humeral distraction while applying inferior glide in the resting position of the glenohumeral joint. Patients had 3 sessions of joint mobilization per week for 6 weeks.
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION
- Group (B) (Experimental): Median nerve mobilization techniques (ULLT-1) in addition to GH joint mobilization
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION

INTERVENTIONS:
Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — Patients were in supine lying position during the whole treatment. The techniques were performed in a rhythmic way, with 2 seconds of glide distraction and then a 2-second break. Each technique was done for 2 minutes [36]. Posterior gliding was performed by maintaining lateral humeral distraction with the glenohumeral in abduction range and the scapula stabilized. Then the therapist applied posterior glide in an oscillating manner. For inferior gliding, with the scapula stabilized, the therapist maintained lateral humeral distraction while applying inferior glide in the resting position of the glenohumeral joint. Patients had 3 sessions of joint mobilization per week for 6 weeks.
  Other Names: joint mobilization
Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — Patients also in this group remained in supine lying position. Median nerve mobilization was performed by placing the scapula in a depressed position with one hand while placing the elbow in 90° flexion, forearm in supination, and wrist and fingers in extension with the other hand. Then, the therapist passively abducted the shoulder into 90- 100° and available external rotation ROM of the arm. Then from this position, the therapist extended the elbow with or without contra lateral side bending of the neck (tensioner or slider technique, respectively). Patients performed 30 repetitions of slider median nerve mobilization by performing elbow extension and wrist extension, with the neck placed in ipsilateral side bending or performing elbow flexion and wrist flexion with the neck placed in contralateral side bending. [35]. Tensioner technique was performed by applying simultaneous elbow extension with contralateral side bending of the neck and hold for 15 sec and relax for 10 sec .
  Arms: Group (B)

SUMMARY:
Background: Adhesive capsulitis (AC) is a common musculoskeletal disorder affecting the functional activities of daily living through capsular restriction. There is a limited knowledge concerning neural restriction as a source of movement limitation in patients with AC other than the enriched knowledge regarding joint mobilization techniques in addressing mobility restrictions for patients with AC. Objectives: This study was designed to determine the efficacy of adding median nerve mobilization to the glenohumeral (GH) joint mobilization techniques on shoulder pain intensity, functional disability and active and passive ROM of glenohumeral abduction and external rotation in patients with AC. Methods: Thirty patients with primary AC with their ages ranged from 40 to 70 years old were included and randomly assigned into two groups. Group A received GH joint mobilization techniques while patients in group B received median nerve mobilization in addition to GH joint mobilization. Both groups received conventional physical therapy which included hot pack for 10 minutes, pendulum exercise and stretching exercises. Treatment sessions were three per week for six weeks. Patients were assessed pre and post interventional procedures for shoulder pain intensity by visual analogue scale (VAS), functional disability by shoulder pain and disability index (SPADI) and active and passive ROM of GH abduction and external rotation by conventional goniometer

DETAILED DESCRIPTION:
Methods:

Study Design: a randomized single blinded controlled trial. This study was conducted at the outpatient clinic of physical therapy, department of rehabilitation and health sciences, college of applied medical sciences, Prince Sattam bin Abdulaziz University over a period from to April to septemper 2024.

Sample size calculation:

Sample size calculation was carried out using g power statistical analysis software (version 3.1.9.2) and revealed that the required size of each group was 26. This calculation was made using α level of 0.05, β=0.2 and large effect size =0.8. Sample size included 20% more than that calculated in anticipation of withdrawal from the experiment (30 in each group). Calculation also based on post treatment data of external ROM measurements from a previous study done by Jung et al

Patients:

Patients were recruited from nearby hospitals and health care facilities and through personal contacts in Al-Kharj city. Ethical approval was granted by the institutional human ethical committee (NO.RHPT/024/007), and patients who agreed to participate signed a written informed consent in accordance with the declaration of Helsinki.

Thirty patients were randomly assigned int 2 groups. Group A(n=15) received oscillatory GH posterior and inferior glide while patients in group B (n=15) received median nerve mobilization (ULLT-1) in addition to GH joint mobilization. All patients in both groups received traditional physical therapy which included hot pack for 10-15 minutes, pendulum exercises and stretching exercises. Patients received three sessions per week for six week and they were evaluated pre and post treatment for shoulder pain intensity by visual analogue scale, functional disability by Shoulder pain and disability index (SPADI) and active and passive ROM of GH abduction and external rotation by conventional goniometer.

Inclusion criteria:

Patients from both genders were included in this study if they would have primary AC with their ages between 40 and 70 years old and complained of pain, stiffness, and limitation of passive shoulder lateral rotation, abduction, and internal rotation of greater than 50%compared to the non-affected side for at least 3 months. Patients with positive (ULTT-1) were also included in this study .

Exclusion criteria:

Patients were excluded if they would have stroke, Parkinson's diseases that interfere with shoulder muscles activity, diabetes, traumatic shoulder conditions, glenohumeral osteoarthritis confirmed by x-ray, previous surgery and manipulation under anesthesia of the affected shoulder [39]. Patients with restricted passive elbow extension ROM were also excluded.

Methods:

Assessment of shoulder pain intensity:

Assessment of shoulder pain intensity was measured by visual analogue scale (VAS) [40] which consists of a horizontal line from 0 to 10 where zero end refers to no pain while the other end refers to great pain. It is a reliable test for literate and illiterate patients 0.94,0.71 respectively) . The patient was asked to mark a point on the line of VAS that represents his or her pain severity. The VAS score was determined by measuring in millimeters from the left-hand end of the line to the point that the patient marked . The obtained score was recorded and was used for statistical analysis .

Assessment of shoulder functional disability:

Shoulder Pain and Disability Index (SPADI) which is a self-questionnaire was used to assess the shoulder pain severity and its influence on functional abilities and activities of daily. Two subscales are included: "Pain" and "Disability". The "Pain" subscale determines the intensity and frequency of glenohumeral pain. In contrast, the "Disability" subscale assesses the impact of pain on activities of daily living, such as self-care, work, and recreational activities. Each subscale involves various factors rated on a Likert scale, where patients experience pain or difficulty. The overall SPADI score was calculated after adding the results of each subscale together. The lowest score is 0 while 100 is the highest score which means that greater grade of pain and functional disability.

Assessment of shoulder ROM:

Conventional goniometer was used to assess active and passive shoulder ROM. It is a highly reliable method (0.94-0.98 test-retest reliability. Patients in this study were assessed for active and passive ROM of glenohumeral abduction and external rotation (with the arm at 0 degrees of abduction) . All Measurements of shoulder ROM were performed three times, and the mean values were used for the statistical analysis

Assessment of GH abduction and external rotation ROM:

For measurement of GH abduction ROM, the patient was in supine lying with shoulder in neutral position; the therapist aligned the fulcrum of the goniometer at the anterior acromial aspect and the movable arm along the anterior aspect of the humerus and the stationary arm was parallel to midline of sternum, the patient was asked to actively elevate his arm in abduction as much as he could, and the reading of the goniometer was noted and was recorded after taking the average of three trials. The passive ROM was performed with the same maneuver but the therapist himself raised the patient's shoulder in abduction through the available range the patient could reach .

For measurement of GH external rotation, the patient was in supine lying with the arm 90 degree abducted and 90-degree elbow flexed. The fulcrum of the goniometer was placed over the olecranon process, the stationary arm was perpendicular to floor, and the movable arm was parallel to the axis ulnar shaft. The patient was asked to actively rotate the arm externally as much as possible, and the reading of the goniometer was noted and was recorded after taking the average of three trials. The passive ROM was performed with the same maneuver but the therapist himself passively rotated the patient's arm externally through the available range the patient could reach

.Interventional procedures: Group (A): GH Joint mobilization techniques (Posterior, Inferior glide). Patients were in supine lying position during the whole treatment. The techniques were performed in a rhythmic way, with 2 seconds of glide distraction and then a 2-second break. Each technique was done for 2 minutes [36]. Posterior gliding was performed by maintaining lateral humeral distraction with the glenohumeral in abduction range and the scapula stabilized. Then the therapist applied posterior glide in an oscillating manner. For inferior gliding, with the scapula stabilized, the therapist maintained lateral humeral distraction while applying inferior glide in the resting position of the glenohumeral joint. Patients had 3 sessions of joint mobilization per week for 6 weeks.

Group (B): Median nerve mobilization techniques (ULLT-1) in addition to GH joint mobilization

Patients also in this group remained in supine lying position. Median nerve mobilization was performed by placing the scapula in a depressed position with one hand while placing the elbow in 90° flexion, forearm in supination, and wrist and fingers in extension with the other hand. Then, the therapist passively abducted the shoulder into 90- 100° and available external rotation ROM of the arm. Then from this position, the therapist extended the elbow with or without contra lateral side bending of the neck (tensioner or slider technique, respectively). Patients performed 30 repetitions of slider median nerve mobilization by performing elbow extension and wrist extension, with the neck placed in ipsilateral side bending or performing elbow flexion and wrist flexion with the neck placed in contralateral side bending. [35]. Tensioner technique was performed by applying simultaneous elbow extension with contralateral side bending of the neck and hold for 15 sec and relax for 10 sec .

Patients in both groups had traditional physical therapy which included 15-20 minutes of hot pack placed under the axilla before mobilization and pendulum exercises to relax and reduce the tension of the glenohumeral muscles . In addition to that, stretching exercises for glenohumeral muscles in the direction of forward elevation, external rotation, horizontal adduction and internal rotation were performed three times per day with holding for 1-5 sec .

Statistical analysis Results were statistically analyzed using SPSS 21, Windows version. All data were expressed as mean ± SD. The Shapiro-Wilk test was used to calculate the normal distribution of scores. For between-group comparison, the independent t-test was used dependent t-test was used for within group comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patients from both genders were included in this study if they would have primary AC with their ages between 40 and 70 years old and complained of pain, stiffness, and limitation of passive shoulder lateral rotation, abduction, and internal rotation of greater than 50%compared to the non-affected side for at least 3 months. Patients with positive (ULTT-1) were also included in this study .

Exclusion Criteria:

* Patients were excluded if they would have stroke, Parkinson's diseases that interfere with shoulder muscles activity, diabetes, traumatic shoulder conditions, glenohumeral osteoarthritis confirmed by x-ray, previous surgery and manipulation under anesthesia of the affected shoulder. Patients with restricted passive elbow extension ROM were also excluded.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
glnohumeral ROM | At baseline and after 6 weeks
  Assessment of shoulder ROM:
  Conventional goniometer was used to assess active and passive shoulder ROM. It is a highly reliable method (0.94-0.98 test-retest reliability. Patients in this study were assessed for active and passive ROM of glenohumeral abduction and external rotation (with the arm at 0 degrees of abduction) . All Measurements of shoulder ROM were performed three times, and the mean values were used for the statistical analysis
  Assessment of GH abduction and external rotation ROM:
  For measurement of GH abduction ROM, the patient was in supine lying with shoulder in neutral position; the therapist aligned the fulcrum of the goniometer at the anterior acromial aspect and the movable arm along the anterior aspect of the humerus and the stationary arm was parallel to midline of sternum, the patient was asked to actively elevate his arm in abduction as much as he could, and the reading of the goniometer was noted and was recorded after taking the average of three trials. T

SECONDARY OUTCOMES:
glenohumeral disability | At baseline and after 6 weeks
  Assessment of shoulder functional disability:
  Shoulder Pain and Disability Index (SPADI) which is a self-questionnaire was used to assess the shoulder pain severity and its influence on functional abilities and activities of daily. Two subscales are included: "Pain" and "Disability". The "Pain" subscale determines the intensity and frequency of glenohumeral pa
glenohumeral pain intensity | At baseline and after 6 weeks
  Assessment of shoulder pain intensity:
  Assessment of shoulder pain intensity was measured by visual analogue scale (VAS) [40] which consists of a horizontal line from 0 to 10 where zero end refers to no pain while the other end refers to great pain. It is a reliable test for literate and illiterate patients 0.94,0.71 respectively) . The patient was asked to mark a point on the line of VAS that represents his or her pain severity. The VAS score was determined by measuring in millimeters from the left-hand end of the line to the point that the patient marked . The obtained score was recorded and was used for statistical analysis .

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Sattam bin Abdulaziz University, Riyadh, Alkharj, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
No need

REFERENCES:
- [Result] Yang JL, Chang CW, Chen SY, Wang SF, Lin JJ. Mobilization techniques in subjects with frozen shoulder syndrome: randomized multiple-treatment trial. Phys Ther. 2007 Oct;87(10):1307-15. doi: 10.2522/ptj.20060295. Epub 2007 Aug 7. PMID 17684085
- [Result] Schmid AB, Brunner F, Luomajoki H, Held U, Bachmann LM, Kunzer S, Coppieters MW. Reliability of clinical tests to evaluate nerve function and mechanosensitivity of the upper limb peripheral nervous system. BMC Musculoskelet Disord. 2009 Jan 21;10:11. doi: 10.1186/1471-2474-10-11. PMID 19154625
- [Result] Akhtar M, Karimi H, Gilani SA, Ahmad A, Raza A. The effectiveness of routine physiotherapy with and without neuromobilization on pain and functional disability in patients with shoulder impingement syndrome; a randomized control clinical trial. BMC Musculoskelet Disord. 2020 Nov 21;21(1):770. doi: 10.1186/s12891-020-03787-0. PMID 33220710
- [Result] Joshi D, Shah S, Shinde SB, Patil S. Effect of Neural Tissue Mobilization on Sensory-Motor Impairments in Breast Cancer Survivors with Lymphedema: An Experimental Study. Asian Pac J Cancer Prev. 2023 Jan 1;24(1):313-319. doi: 10.31557/APJCP.2023.24.1.313. PMID 36708582
- [Derived] Hegazy MMA, Mahmoud WSE, Ahmed AS. Slider Versus Tensioner Median Nerve Mobilization in Patients With Frozen Shoulder Randomized Controlled Comparative Study. Physiother Res Int. 2026 Jan;31(1):e70164. doi: 10.1002/pri.70164. PMID 41549328